CLINICAL TRIAL: NCT02752789
Title: An Observational Cohort Study to Determine the Impact of Alloantibodies and Antibodies to Self Antigens on Chronic Graft Function up to 5 Years After Pediatric Heart Transplantation (CTOTC-09)
Brief Title: Impact of Allo- and Autoantibodies on Chronic Cardiac Allograft Function
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation in Children (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOTC-09
Record Dates: First submitted 2016-04-22; First posted 2016-04-27 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Pediatric Heart Transplantation; Pediatric Heart Transplant Recipients
Keywords: alloantibodies; donor specific antibodies (DSA)-preformed, de novo; self-antigens; chronic allograft function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, PBMC and tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pediatric Heart Transplant Recipients: CTOTC-04 (ClinicalTrials.gov ID NCT01005316) participants who consent to long-term follow-up as part of this study as well as candidates less than 21 years of age who are listed for isolated orthotopic heart transplantation at one of the participating sites

SUMMARY:
This is a multi-center, prospective, single cohort, observational study of pediatric heart transplant recipients designed to determine the impact of preformed versus de novo human leukocyte antigen (HLA) donor-specific antibodies (DSA), and antibodies to the self-antigens cardiac myosin and vimentin, on chronic allograft function. In addition, the investigators will explore mechanisms of action and predictors of DSA, rejection and altered pathophysiology.

DETAILED DESCRIPTION:
Participants that were enrolled in the CTOTC-04 study (ClinicalTrials.gov Identifier NCT01005316) are invited to enroll in this CTOTC-09 study. Conversion from the CTOTC-04 to CTOTC-09 study will occur in such a manner as to avoid/minimize discontinuity of follow-up between the planned CTOTC-04 and CTOTC-09 study visits. In addition, subjects added to the United Network for Organ Sharing (UNOS) system-or Canadian equivalent agency-at a participating study site, who are less than 21 years of age and fulfill all study eligibility criteria, will be invited to enroll in CTOTC-09.

This study focuses on the importance of antibodies against the newly transplanted heart in pediatric heart transplant recipients. The investigators aim to determine if certain antibodies lead to problems with the heart transplant. Antibodies are small proteins in the blood that the body makes to fight off infections, for example with bacteria or viruses. Since a new heart is "foreign" to the recipient's body, their immune system might try to attack it with antibodies, as if it were an infection. For many years it was thought that only white blood cells attacked the new heart, causing rejection.

Now there is new information showing that antibodies may also cause rejection or long-term damage to the heart. At this time, very little is known about how antibodies might cause problems after heart transplantation in transplant recipients younger than 21 years at the time of transplant.

This study will collect a medical history and blood samples at specified times for research. The blood samples will be used to measure antibodies in the blood, and to perform special tests to see how these antibodies might damage the heart.

Participant follow-up is from the day of the heart transplant to year 5 post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or parent guardian able to understand and provide informed consent and where applicable assent
* Planned long-term follow-up at one of the study sites

AND either:

-Enrolled in the CTOTC-04 study and actively followed at one of the study sites

OR

-Listed at participating study sites, less than 21 years of age and not yet transplanted.

The inclusion criteria for enrollment of new study patients in the CTOTC-09 Protocol will be the same as the CTOTC-04 study (refer to ClinicalTrials.gov ID NCT01005316).

Exclusion Criteria:

* Parental withdrawal of consent from the CTOTC-04 study
* Past or current medical problems or findings from physical examination or laboratory testing that, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or may impact the quality or interpretation of the data obtained from the study
* Listed for simultaneous multiple organ transplant.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants that were enrolled in CTOTC-04 (ClinicalTrials.gov ID NCT01005316) who consent to long-term follow-up and new participants at the nine designated sites who are listed for isolated orthotopic heart transplantation
Sampling Method: Non-Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary capillary wedge pressure at heart catheterization | 3 years post-transplantation

SECONDARY OUTCOMES:
Other invasive cardiac hemodynamic findings at cardiac catheterization | 3 and 5 years post-transplantation
  Cardiac hemodynamic findings: right and left ventricular end diastolic pressures, right atrial pressure, pulmonary artery pressure and cardiac index
Frequency of development of post-transplant de novo DSA and autoantibodies to cardiac myosin and vimentin | 3 years post-transplantation
Time course of development of post-transplant de novo DSA and autoantibodies to cardiac myosin and vimentin. | 3 years post-transplantation
Frequency of first episode of late acute rejection | From >1 year to 5 years post-transplantation
Time to first episode of late acute rejection | From >1 year to 5 years post-transplantation
  Late acute rejection is defined as occurring >1 year post-transplantation
Frequency to recurrent (two or more) late acute rejections | Up to 5 years post-transplantation
Time to recurrent late acute rejections | Up to 5 years post-transplantation
  Recurrent defined as two or more late acute rejection episodes
Frequency to first episode of late acute rejection with hemodynamic compromise | Up to 5 years post-transplantation
Time to first episode of late acute rejection with hemodynamic compromise | Up to 5 years post-transplantation
Time to graft loss (death or retransplantation) conditional to surviving one year post-transplantation | One year and up to 5 years post-transplantation
N-terminal pro-brain Natriuretic Peptide (NT-proBNP)/Brain Natriuretic Peptide (BNP) | 3 and 5 years post-transplantation
Systolic and diastolic graft function | 3 and 5 years
  Graft function as assessed by echocardiography
Proportion of participants with angiographic evidence of coronary artery disease | 3 and 5 years post-transplantation
Time to graft loss (death or retransplantation) after first late rejection | Up to 5 years post-transplantation
Medication Adherence Measure (MAM) after hospital discharge | Up to 5 years post-transplantation
Variability of maintenance tacrolimus levels | Up to 5 years post-transplantation

OTHER OUTCOMES:
Exploratory: Microvascular pathology | Up to 5 years post-transplantation
  Microvascular pathology as defined by:
  * cytoprotective intracellular signaling (bcl2, Heme Oxygenase-1(HO-1))
  * interstitial capillary network
  * endothelial cell progenitor influx and premature senescence
  * obliterative microvasculopathy (arteriolopathy)
Exploratory: Expression of cytoprotective genes Bcl2 and HO-1, ICAM, VCAM and selectins, Complement inhibitory proteins CD55, CD59, CR1, CR2 and CR3. | After exposure to alloantibody (or control) (At Year 1)
  Endothelial Cell (EC) Culture Model is used to study factors that will predict and contribute to the protection of the graft following transplantation across sub-threshold concentrations of DSA. Exploratory: Expression of cytoprotective genes Bcl2 and HO-1, Intercellular adhesion molecules (ICAM), Vascular Cell Adhesion Molecule (VCAM) and selectins, Complement inhibitory proteins (cluster of differentiation antigen 55 (CD55), cluster of differentiation antigen 59 (CD59), Complement Receptor 1 (CR1), (CR2) and (CR3).
Exploratory: Cellular immune responses to allo-antigens and self-antigens (vimentin and myosin) | 24 hours prior transplantation, Months 3 and 6 post transplantation
  Cellular immune responses to allo-antigens and self-antigens (vimentin and myosin) will be measured by:
  * ELISPOT for Interleukin 17 (IL17) and Interleukin 10 (IL10) producing T cells
  * Plasma cytokines by Luminex (IL-6, IL-1beta, IL-17, Cxcl12, IL-10 and Transforming Growth Factor-beta (TGF-beta)
Exploratory: Role of Interleukin-33 (IL-33) and its Receptor (ST2) in cardioprotection against effects of DSA | Month 5 post transplantation
  Role of IL-33 and its Receptor (ST2) in cardioprotection against effects of DSA will be measured by:
  * IL33 and ST2 expression in graft biopsies
  * Soluble ST2 in serum

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Webber, MBChB, MRCP, Study Chair — Monroe Carell Jr. Children's Hospital at Vanderbilt: Pediatric Transplantation; Steven A. Webber, MBChB, MRCP, Principal Investigator — Monroe Carell Jr. Children's Hospital at Vanderbilt: Pediatric Transplantation
Locations (9):
- United States (8):
  - Emory University School of Medicine, Atlanta, Georgia
  - Children's Hospital Boston, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Children's Hospital at Montefiore, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital, Nashville, Tennessee
- Hospital for Sick Children, Toronto, Canada

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Clinical Trials in Organ Transplantation in Children (CTOT-C) — http://www.ctotc.org/